CLINICAL TRIAL: NCT04119271
Title: Durham Healthy Breathing in Healthy Homes Project: A Duke-Reinvestment Partners Collaborative
Brief Title: Durham Healthy Breathing in Healthy Homes Project
Acronym: DHBHH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Reinvestment Partners (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00102762
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-02

CONDITIONS: Poor Asthma Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breathe Easy at Home Kit Products (Other): Families will be provided with a Breathe Easy at Home Kit. These kits will include:
  a HEPA filtered upright vacuum cleaner, a HEPA-filtered Air Purifier, a Hypoallergenic latex free mattress cover, box spring cover, and two pillow covers, Healthier alternative to most household cleaners, Non- toxic glue type pest control devices for rodent control, and a combination of safe products to locate and kill roaches.
  Interventions: Other: Breathe Easy at Home Kit Products

INTERVENTIONS:
Other: Breathe Easy at Home Kit Products — HEPA filtered upright vacuum cleaner, HEPA-filtered Air Purifier, Hypoallergenic latex free mattress cover, box spring cover, and two pillow covers, Healthier alternative to most household cleaners, Non- toxic glue type pest control devices for rodent control and a combination of safe products to locate and kill roaches.

SUMMARY:
To determine if Home-based Environmental Interventions (HEI) that improve home air-quality problems can improve asthma outcomes. Participants will benefit through home-based environmental interventions that improve home air-quality problems and improve asthma outcomes. All participants will receive a Breath Easy at Home Kit, which could help with reducing environmental exposures. The primary objective is to assess the feasibility and acceptability of the HEI measured by the proportion of families completing intervention components and proportion of caregivers expressing satisfaction with intervention components. Secondary objective is to explore the efficacy of a HEI on reducing environmental exposures measured using personal wristband monitors.

Exploratory objective is improvements in asthma control following HEI measured using asthma control scores and lung function. The fourth objection is to explore correlations between demographics, body weight, housing characteristics (smokers, electronic cigarette use, number of pets, housing type) with measures of acceptability, satisfaction and improved exposure markers.

DETAILED DESCRIPTION:
The investigator propses a 23-week prospective, open label, single center, environmental remediation intervention study in 5-16 year old children with poor asthma control. At visit 1, wristbands will be dispensed and collected to estimate exposure to a suite of common organic contaminants including phthalates, organophosphate esters, several pesticides and polyaromatic hydrocarbons (PAH). During the initial home visit, the Healthy Homes Housing Specialist will conduct an environmental home assessment to identify asthma triggers in accordance with the EPA's recommendations for helping children with asthma. The Housing Specialist will follow the EPA document Home Characteristics and Asthma Triggers, and will provide the family with a Breathe Easy at Home Kit. The Specialist will provide training and instructions on how to use each of the supplies provided in the kit. If the Housing Specialist identifies necessary home repairs during the assessment process, the Housing Specialist can refer the family to organizations that offer home repairs, modifications, and weatherization services. The specialist will discuss the importance of clean air for maintaining lung health for all family members and will discuss the importance of banning of any indoor smoking, smoking anywhere around the household and smoking in any household automobiles (even when the child is not present). Follow up phone calls will be conducted to answer questions, complete questionnaires and complete a household environmental interview.

ELIGIBILITY:
Inclusion Criteria:

* Parent/legal guardian has provided informed consent (child has provided assent if needed)
* 5-16 years of age with physician-diagnosed asthma
* Evidence of poor asthma control defined as either:

Hospitalization at Duke Children's Hospital within past 30 days or, ACQ6 > 1.0 during ambulatory visit to Duke Asthma Center within 2 weeks

Exclusion Criteria:

* Lack of informed consent
* Any major chronic illness that in the opinion of the PI would interfere with participation in the intervention or completion of the study procedures
* Inability to complete baseline measurements in a satisfactory manner according to the judgment of the research coordinator or PI
* Family is planning to move households in the next 2 months
* Parent/Caregiver unable to consent in English
* Sensitivity or allergy to silicone

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Number of completed home visits as measured by completion logs | 2 months
Number of completion of the post-intervention phone visit as measured by call logs | Four Months
Number of caregiver reporting satisfaction with intervention as measured by survey responses | Four Month

SECONDARY OUTCOMES:
Change in Environmental Wristband Markers | 3 weeks and 7 weeks
  changes in targeted environmental wristband markers of exposure to organic contaminants in the home environment, including phthalates, organophosphate esters, several pesticides, and polyaromatic hydrocarbon (PAH) markers evaluated using personal silicone wristband monitors. Paired t-tests (or Wilcoxon signed rank tests for non-parametric data) will be used to assess post-intervention changes in targeted wristbands toxin levels.The relationship between changes in these outcomes and measures of intervention adherence will be analyzed using Pearson correlations and ANOVA trend testing as appropriate.
Change in Indoor Air Quality measured by questionnaire | 3 weeks and 7 weeks
  Sponsor developed questionnaire-15 to 20 questions asking about air quality.
Change in Asthma Symptoms | 1 week and 4 months
  Change in asthma symptom control measured by the asthma control questionnaire 6 (ACQ6) (ambulatory participants only).
Change in Spirometry Values as measured by spirometric measures | 1 week and 4 months
  Impulse Oscillometry (IOS) simply requires the child to breathe in and out through a mouthpiece for 20-30 seconds. During breathing, a loudspeaker delivers a quiet pulse-shaped pressure-flow signal to the respiratory system. Spirometric measures is the forced vital capacity (FVC),
Change in Asthma Symptoms | 1 week and 4 months
  Improvements in asthma control following HEI measured using asthma control scores and lung function. For patients enrolled in the ambulatory setting, change in FEV1, FEV1/FVC by spirometry will be calculated.
Change in Spirometry Values as measured by spirometric measures | 1 week and 4 months
  The Spirometer measure is theforced expiratory volume in 1 second (FEV1),
Change in Spirometry Values as measured by spirometric measures | 1 week and 4 months
  The Spirometeric Measure is the FEV1/FVC ratio
Change in Spirometry Values as measured by spirometric measures | 1 week and 4 months
  The Spirometric Measure is the forced expiratory flow average over 25-75% of FVC (FEF25-75).

CONTACTS AND LOCATIONS:
Overall Officials: Jason E Lang, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No